CLINICAL TRIAL: NCT07114029
Title: Anatomic and Functional Comparison of Preoperative and Postoperative Outcomes of Mesh Free Sacrocolpopexy Performed Via Vaginal Natural Orifice Transluminal Endoscopic Surgery (VNOTES)
Brief Title: VNOTES Approach in Mesh Free Sacrocolpopexy: A Functional and Anatomic Evaluation
Acronym: vnotes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: gopvnotes
Record Dates: First submitted 2025-07-10; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: sacrocolpopexy; mesh-free
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, single-center interventional study designed to evaluate the anatomical and functional outcomes of mesh-free sacrocolpopexy performed via the VNOTES technique in patients with pelvic organ prolapse. All participants will undergo the same surgical intervention without randomization or a comparator arm. Preoperative and postoperative evaluations will be conducted using standardized tools over a 6-month follow-up period. The study is open-label, with no masking applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesh-free Sacrocolpopexy via VNOTES (Experimental): Mesh-free sacrocolpopexy is performed via the VNOTES technique to treat pelvic organ prolapse. Outcomes will be evaluated before and 6 months after surgery.
  Interventions: Procedure: Mesh-free Sacrocolpopexy via VNOTES

INTERVENTIONS:
Procedure: Mesh-free Sacrocolpopexy via VNOTES — Mesh-free sacrocolpopexy is performed via the VNOTES technique to treat pelvic organ prolapse. Outcomes will be evaluated before and 6 months after surgery.

SUMMARY:
This study aims to evaluate the effectiveness of mesh-free sacrocolpopexy performed using the VNOTES (Vaginal Natural Orifice Transluminal Endoscopic Surgery) technique in the surgical treatment of pelvic organ prolapse. Anatomical and functional outcomes will be assessed over a 6-month period before and after the operation. Evaluation tools will include the Pelvic Floor Distress Inventory-20 (PFDI-20), Pelvic Organ Prolapse Quantification (POP-Q) system, and the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12).

The findings of this study are expected to provide important data on the anatomical improvement, functional outcomes, and impact on sexual function of mesh-free sacrocolpopexy performed via the VNOTES approach.

DETAILED DESCRIPTION:
This prospective clinical study investigates the anatomical and functional outcomes of mesh-free sacrocolpopexy performed using the VNOTES (Vaginal Natural Orifice Transluminal Endoscopic Surgery) technique in the surgical treatment of pelvic organ prolapse. The VNOTES approach allows transvaginal access to the pelvic cavity without the need for abdominal incisions, offering the advantages of minimally invasive surgery while avoiding the use of synthetic mesh.

The study includes women diagnosed with stage II or higher pelvic organ prolapse who are candidates for sacrocolpopexy via the VNOTES technique. All participants will undergo mesh-free sacrocolpopexy performed transvaginally using endoscopic guidance.

Anatomical and functional outcomes will be evaluated using validated tools, including the Pelvic Organ Prolapse Quantification (POP-Q) system, the Pelvic Floor Distress Inventory-20 (PFDI-20), and the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Assessments will be performed preoperatively and at 6 months postoperatively. Intraoperative data such as operative time, estimated blood loss, complications, and length of hospital stay will also be collected.

The primary goal of the study is to assess anatomical success based on changes in POP-Q staging. Secondary outcomes include improvements in pelvic floor symptoms, sexual function, recurrence rates, and patient satisfaction.

This study aims to provide evidence on the safety, feasibility, and functional benefits of performing sacrocolpopexy without mesh through the VNOTES approach in the management of advanced pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

Patients who applied to Gaziosmanpasa Education and Research Hospital, Gynecology and Obstetrics Clinic, have apical and anterior POP Q stage 2 and above, and have undergone surgery due to symptomatic pelvic organ prolapse, Patients who are over the age of 18 and who are citizens of the Republic of Turkey, and who have undergone surgery by experienced surgeons will be included in the study.

Exclusion Criteria:

Having previously received KT and/or RT due to any malignancy Having previously undergone surgery due to prolapse Patients with severe cardiovascular or respiratory diseases will not be included in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory-20 (PFDI-20) Score Change | Baseline to 6 months postoperative
  Change in pelvic floor symptom distress measured by PFDI-20 questionnaire.
Pelvic Organ Prolapse Quantification (POP-Q) Score Change | Baseline to 6 months postoperative
  Change in anatomical prolapse stage evaluated by POP-Q scoring system.
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) Score Change | Baseline to 6 months postoperative
  Change in sexual function assessed by PISQ-12 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: süleyman salman, professor, Study Director — Gaziosmanpasa Training and Research Hospital; havva betül bacak, md, Principal Investigator — Gaziosmanpasa Training and Research Hospital
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No